CLINICAL TRIAL: NCT05319938
Title: Clinical Evaluation of Treatment With Micro-surgical Management of Type I Multiple Gingival Recessions Using Coronally Advanced Flap With Either Advanced Platelet-Rich Fibrin or Concentrated Growth Factor: A Comparative Analysis
Brief Title: Growth Factors in the Treatment of the Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen Öngöz Dede, Clinical Association Professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD-1726
Record Dates: First submitted 2022-03-11; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Growth Factors, Combined Defect of; Gingival Recession
MeSH Terms: conditions — Growth Factors, Combined Defect of; Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAF only (Active Comparator): Only Coronally Advanced Flap technique
  Interventions: Procedure: CAF only
- CAF+CGF (Experimental): Concentrated Growth Factor (CGF) applied together with Coronally Advanced Flap (CAF) technique
  Interventions: Procedure: CAF+CGF
- CAF+A-PRF (Experimental): Advanced Platelet-Rich Fibrin (A-PRF) applied together with Coronally Advanced Flap (CAF) technique
  Interventions: Procedure: CAF+A-PRF

INTERVENTIONS:
Procedure: CAF only — After local anesthesia, initially, sulcular incisions were made on the buccal aspect of the teeth and two vertical incisions were made. A trapezoidal flap was elevated with a split-full-split approach in the coronal-apical direction. The anatomic inter-dental papillae adjacent to the involved tooth were de-epithelialized. Plaque, calculus, and soft tooth structures on exposed root surfaces were removed with curettes. No further mechanical or chemical root conditioning materials were performed. The flap was coronally placed over the membranes to completely cover the CEJ and sutured with 6.0 propylene suture.
  Arms: CAF only
Procedure: CAF+CGF — After local anesthesia, initially, sulcular incisions were made on the buccal aspect of the teeth and two vertical incisions were made. A trapezoidal flap was elevated with a split-full-split approach in the coronal-apical direction. The anatomic inter-dental papillae adjacent to the involved tooth were de-epithelialized. Plaque, calculus, and soft tooth structures on exposed root surfaces were removed with curettes. No further mechanical or chemical root conditioning materials were performed. The flap was coronally placed over the membranes to completely cover the CEJ and sutured with 6.0 propylene suture.
  Blood samples were collected into 10 ml glass-coated plastic tubes without anticoagulant solutions. These tubes were placed into CGF centrifuge machine and centrifuged immediately . CGF membrane were placed over the defect. The flap was coronally placed over the membranes to completely cover the CEJ and sutured with 6.0 propylene suture.
  Arms: CAF+CGF
Procedure: CAF+A-PRF — After local anesthesia, initially, sulcular incisions were made on the buccal aspect of the teeth and two vertical incisions were made. A trapezoidal flap was elevated with a split-full-split approach in the coronal-apical direction. The anatomic inter-dental papillae adjacent to the involved tooth were de-epithelialized. Plaque, calculus, and soft tooth structures on exposed root surfaces were removed with curettes. No further mechanical or chemical root conditioning materials were performed. The flap was coronally placed over the membranes to completely cover the CEJ and sutured with 6.0 propylene suture.
  Blood samples were collected into 10 ml glass-coated plastic tubes without anticoagulant solutions. These tubes were placed into A-PRF centrifuge machine and centrifuged immediately. A-PRF membrane were placed over the defect. The flap was coronally placed over the membranes to completely cover the CEJ and sutured with 6.0 propylene suture.
  Arms: CAF+A-PRF

SUMMARY:
The purpose of this study was to compare and evaluate the clinical effects of Concentrated Growth Factor (CGF) and Advanced Platelet-Rich Fibrin (A-PRF) applied together with Coronally Advanced Flap (CAF) technique using a microsurgical approach in the treatment of Type I multiple gingival recessions (GR).

ELIGIBILITY:
Inclusion Criteria:

* Systematically and periodontally healthy non-smokers
* Presence of Cairo Recession type I gingival recession with ≥ 2 mm gingival recession depth, probing depth <3 mm and gingival thickness (GT) ≥ 0.8 mm on both sides of the maxillary arch
* Width of keratinized gingiva ≥ 2mm
* Presence of identifiable cemento-enamel junction
* Full-mouth plaque index (PI) < 20 %
* Gingival index (GI) scores =1
* Presence of tooth vitality
* Absence of caries, restorations and furcation involvement in the treated area

Exclusion Criteria:

* Patients who had systemic problems that wound contraindicate for periodontal surgery
* Usage of medications known to interfere with healing and to cause gingival enlargement
* Recession defects associated with demineralization, deep abrasion, previous surgery in the defects area within the past 1 year
* Pregnant or lactating females
* Drug and alcohol abuse

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Complete and mean root coverage | Change from baseline at 6 months of the percent of complete and mean root coverage
  Percentages of root coverage and complete root coverage were calculated according to the following standard formulae.
  Percentage of root coverage: [(preop. vertical gingival recession (VGR)- postop.VGR)\ preop. VGR] x 100 Percentage of complete root coverage: [(teeth with complete root coverage) \ (all treated teeth)] x 100.

SECONDARY OUTCOMES:
Gingival thickness | Change from baseline at 6 months of the gingival thickness
  The gingival thickness was evaluated midbuccally in the attached gingival (GT-MB), halfway between the mucogingival junction and free gingival groove and at the base of the interdental papilla. GT was measured by using a periodontal probe with a rubber stopper under local anesthesia, and then the thickness was assessed by transferring to an electronic digital caliper.
Keratinized gingiva width (WKG) | Change from baseline at 6 months of keratinized gingiva width
  The WKG was determined by subtracting the VGR from the CEJ- MGJ (mucogingival junction).
Patient esthetic score (PES) | Change from baseline at 6 months of the patient esthetic score
  Patient esthetic score (PES) to evaluate esthetic appearance (color, appearance, and form of the selected site),
  PES: bad-unlikely esthetics (score 0) → perfect esthetics (score 10)
Patient comfort score (PCS) | Change from baseline at 6 months of the patient comfort score
  Patient comfort score (PCS) for the pain, edema and other experiences regarding operating technique, instruments, and microscopic view, etc.
  PCS: unbearable discomfort (score 0) → no-discomfort (score 10).
Hypersensitivity score (HS) | Change from baseline at 6 months of the hypersensitivity score
  "Hypersensitivity" score was recorded after blasting air (60 psi, 22°C) derived from a dental syringe that was heading for the root surface for 1 s. The syringe was held at 90° angle, 2-3 mm from the root surface. Neighboring teeth were shielded during testing with the dentist's gloved fingers; then the patient has enquired again to score the discomfort level.
  HS: no pain (score 0) → worst pain imaginable (score 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Figen Öngöz Dede, Ordu, Turkey (Türkiye)